CLINICAL TRIAL: NCT05570578
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Brain Organization and Naming
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Brain Organization and Naming in Aphasic Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adrian Guggisberg (Other)
Responsible Party: Sponsor-Investigator, Adrian Guggisberg, Médecin conseil, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-D0058
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Aphasia
Keywords: tDCS; Functional connectivity; EEG
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: sham-tDCS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD-tDCS (Active Comparator): high-density transcranial direct current stimulation (HD-tDCS) over Broca's area
  Interventions: Device: HD-tDCS
- sham-tDCS (Sham Comparator): sham transcranial direct current stimulation. The same setup will be used as in the HD-tDCS arm, except that the current will be ramped up for 30 seconds and then switched off. This does not lead to neural effects, but the patients have a similar sensation.
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — The anode electrode will be placed over Broca's area, 4 cathode electrodes will be placed at about 2 cm distance each from the anode in 4 directions.
  Other Names: high-density transcranial direct current stimulation; DC-stimulator

SUMMARY:
High-Definition Transcranial Direct Current Stimulation (HD-tDCS) allows to induce, in a non-invasive way, a transient inhibitory or excitatory neuromodulation of a given cerebral region and to obtain a very focused cortical effect. Previous studies using HD-tDCS have shown the effectiveness of this stimulation technique for enhancing language recovery in patients with aphasia.

However, language processes are not determined solely by local neural activity at a single site, but rather by the interaction between neural networks. This is because a large cortical network is involved in language processes and, therefore, the same language disorder may result from lesions at different locations in this network.

The investigators hypothesize that anodal HD-tDCS will enhance neural interactions between language areas and, thereby, improve language processing and word learning.

The investigators propose to carry out a study on chronic aphasic patients involving HD-tDCS of the Broca region (left inferior frontal gyrus) combined with a verb learning task.

DETAILED DESCRIPTION:
Functional connectivity (FC) represents a means of analyzing functional interactions in the brain network by assessing the statistical dependence of neural activity between brain areas. The brain maintains a high level of interactions between brain areas even in the resting state, when it is not explicitly involved in a specific task. Resting-state interactions occur mainly in the so-called alpha frequency band (8-13 Hz) . Moreover, these resting-state interactions are crucial for correct task performance and learning. Indeed, healthy subjects with high resting-state alpha-band FC levels are better able to perform tasks and learn. For example, subjects with high levels of FC between Broca's area and the rest of the brain perform better on language production tasks and show greater training gains when learning new words. In addition, patients with brain damage due to stroke show a reduction in resting-state alpha-band FC, which correlates with the severity of neurological deficits. In particular, a loss of FC of structurally preserved inferior frontal areas was associated with more severe aphasia. Conversely, high-levels of FC between the inferior frontal brain areas and the rest of the brain during the first weeks after stroke was associated with better recovery from aphasia, probably reflecting a reorganization of neural connections as a neural mechanism involved in plasticity. Resting-state FC is therefore an interesting neural target for therapy, which could help improve recovery from aphasia.

In a previous study on healthy subjects, the investigators have indeed observed that HD-tDCS applied to Broca's area improves the ability for new-verb learning, i.e., the correct naming of action pictures. This improvement in learning correlated with greater increase in FC between Broca's and Wernicke's area.

The investigators now carry out a study on chronic aphasic patients involving HD-tDCS of the Broca region (left inferior frontal gyrus) combined with a verb learning task.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke
* Presence of aphasia with difficulty finding words and/or naming objects/pictures
* ≥12 months post-stroke
* ≥ 18 years of age
* French-speaking
* Able to participate in 30-60 min therapeutic sessions (good concentration and understanding of the task and ability to follow instructions

Exclusion Criteria:

* Patients unable to understand the given information on the study and its objectives, or instructions for tasks performed.
* Impaired alertness or delirium
* Severe co-morbidity affecting speech
* Contraindication to tDCS: pregnant women, patients with active implants such as pacemakers or cochlear implants, patients with one or more seizures, metal objects in the brain
* Occurrence of a new stroke during the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Action picture naming, short-term improvement | Change from day 1 (baseline) to day 5 (posttest)
  Change in number of correctly named action pictures

SECONDARY OUTCOMES:
Functional connectivity between Broca's and Wernicke's area | Change from day 1 (baseline) to day 5 (posttest)
  Change in the normalized imaginary component of coherence between Broca and Wernicke

OTHER OUTCOMES:
Action picture naming, long-term improvement | Change from day 1 (baseline) to week 4 (follow-up)
  Change in number of correctly named action pictures
Narrative speech, short-term improvement | Change from day 1 (baseline) to day 5 (posttest)
  Patient describes cookie-theft picture and action-picture, change in score
Narrative speech, long-term improvement | Change from day 1 (baseline) to week 4 (follow-up)
  Patient describes cookie-theft picture and action-picture, change in score

CONTACTS AND LOCATIONS:
Overall Officials: Adrian G Guggisberg, MD, Principal Investigator — University of Geneva
Locations (1):
- Division of Neurorehabilitation, University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Published and analyzed data will be archived in a secure location on a data sharing server that meets the FAIR (Findability, Accessibility, Interoperability, and Reuse) principles for a minimum of 10 years.
Time Frame: Once the study has been published
Access Criteria: Open Access